CLINICAL TRIAL: NCT07203560
Title: Neurodynamic Mobilization for the Management of Patients With Lumbar Disc Herniation: A Randomized Controlled Study
Brief Title: Effect of Neurodynamic Mobilization in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gurkan Gunaydin, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-FTR-GG-01
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Herniation; Low Back Pain
Keywords: low back pain; sciatica; Disability Evaluation; Musculoskeletal Manipulations
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Sciatica

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group randomized controlled trial. Control group received a conventional physiotherapy program; intervention group received the same program plus neurodynamic mobilization. Treatments were delivered over 4 consecutive weeks. Outcomes included pain, ROM, neurodynamic mobility, functional status and disability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodynamic Mobilization + Conventional Therapy (Experimental Group) (Experimental): Participants received the conventional physiotherapy program plus neurodynamic mobilization administered by a physical therapist. Treatment was given 5 days a week for 4 weeks, for a total of 20 sessions.
  Interventions: Other: Neurodynamic Mobilization; Other: Conventional Physiotherapy
- Conventional Therapy (Control Group) (Active Comparator): Individuals in control group received hot therapy (Hotpack, 20 minutes), Conventional Tens (60 Hz, 60 msec, 20 minutes) and Therapeutic Ultrasound (1.5 w/cm2, 10 minutes). Patients were given an exercise program to do at home and the treatment was given 5 days a week for 4 weeks, for a total of 20 sessions, to all patients in the study.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Neurodynamic Mobilization — In the experimental group, neurodynamic mobilization was applied in addition to the conventional physiotherapy program. For the neurodynamic mobilization tibial nerve neural mobilization was performed. For neural mobilization of the tibial nerve, the patient was placed in the side-lying position with the hip in 90° flexion, knee flexion and ankle dorsi flexion. In this position, the ankle and hip positions were maintained, and knee extension was performed. When the symptoms were at a level that would not disturb the patient, it was held for 5 seconds, and knee flexion was performed by plantar flexion of the ankle. This practice was performed twice a week with 10 repetitions by a physiotherapist. The same neurodynamic mobilization exercise was recommended to the patients in the neuromobilization group as a home program with 10 repetitions twice a day.
  Arms: Neurodynamic Mobilization + Conventional Therapy (Experimental Group)
Other: Conventional Physiotherapy — All participants received hot pack therapy (20 minutes), conventional TENS (60 Hz, 60 msec, 20 minutes), therapeutic ultrasound (1.5 W/cm², 10 minutes), and a prescribed home exercise program, delivered 5 days per week for 4 weeks (20 sessions in total).

SUMMARY:
The objective of this randomized controlled trial was to investigate the effects of neurodynamic mobilization on pain intensity, normal joint motion, neurodynamics, functional level, and disability in patients with lumbar disc herniation.

DETAILED DESCRIPTION:
Background: Low back pain is a major cause of disability worldwide, and due to the limited effectiveness of current treatments, this study aimed to evaluate the efficacy of neurodynamic mobilization technique on pain intensity, range of motion, neurodynamics, functional status, and disability in patients.

Methods: Thirty-seven patients were randomized to control or mobilization group. Participants in the control group received a conventional therapy for 20 treatment sessions, and those in the mobilization group were treated neurodynamic mobilization in addition to the electro/thermal therapy program twice a week for 4 consecutive weeks. Pain level at rest and during activity was recorded with a Visual Analog Scale. Active lumbar flexion, extension, and lateral flexion were measured with a universal goniometer. Neurodynamic mobility was evaluated using neurodynamic tests. The functional status was assessed with the 30-second chair stand test and disability was evaluated with the Bournemouth Questionnaire. 2x2 repeated measures ANOVA models were used to determine within and between group differences.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* Diagnosed with lumbar disc herniation at one or more of the L3-L4, L4-L5
* L5-S1 levels with prolapsed, protruding, or extruding disc confirmed by MRI
* Presence of low back pain for at least 6 weeks.

Exclusion Criteria:

* Spinal stenosis
* Previous lumbar surgery or medical treatment for disc herniation
* Pregnancy
* Severe osteoporosis
* Diabetes mellitus
* Severe neurological deficit

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pain was assessed at baseline (before treatment) and at the end of 4 weeks of treatment (post-treatment)
  Patients' rest and activity pain levels was assessed via a visual analog scale (VAS). Participants were asked to mark the intensity of pain they felt on a 10-centimeter (cm) horizontal line (0 indicates no pain, 10 indicates intolerable pain). The point marked on the line was measured with a ruler and the VAS value was recorded in cm

SECONDARY OUTCOMES:
ROM | Rom was assessed at baseline (before treatment) and at the end of 4 weeks of treatment (post-treatment).
  Rom of the lumbar region was evaluated using a universal goniometer. Lumbar flexion and extension, right and left lateral trunk flexion were measured actively and recorded in terms of degree.
Neurodynamic Mobility - Slump Test | These were assessed at baseline (before treatment) and at the end of 4 weeks of treatment (post-treatment).
  Slump test The patient was asked to sit on the edge of the examination table with the knee flexed at 90° and to flex the neck, back, and lower back respectively. He was then asked to bring his big toe towards his head by extending the knee. In this position, the angle between the starting position and the fibula was measured with a universal goniometer. The test was repeated twice and the mean degree was recorded.
Neurodynamic Mobility - Sit and Reach Test | Baseline (before treatment) and at the end of 4 weeks of treatment (post-treatment)
  Sit and Reach test The top of a table with a height of 32 cm and a length of 35 cm was scaled by dividing it into cm. The patient was asked to sit on the floor and rest the sole of her bare foot flat on the test table. She was then instructed to reach as far as possible forward on the table without bending her knees from her trunk. The extreme point at which her fingers extended was measured in cm. In this way, at the farthest point, they waited 1-2 seconds without stretching forward or backward. The test was repeated twice, and the mean was recorded in cm

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Gunaydin, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Gazi University Department of Physical Therapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No